CLINICAL TRIAL: NCT00455650
Title: Cognitive Effects of Mecamylamine and Varenicline in Schizophrenia
Brief Title: Study of the Effects of Mecamylamine and Varenicline in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); The Bowman Family Foundation (Unknown)
Responsible Party: Principal Investigator, A. Eden Evins, Director of Center for Addiction Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC #2006-P-001361; CORRC#3-2007
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Cognition in Schizophrenia
Keywords: schizophrenia; cognition; nicotinic receptors; mecamylamine; varenicline
MeSH Terms: conditions — Schizophrenia | interventions — Mecamylamine; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Schizophrenia, Mecamylamine (Active Comparator)
  Interventions: Drug: Mecamylamine
- Schizophrenia, Varenicline (Active Comparator)
  Interventions: Drug: Varenicline
- Schizophrenia, Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Control, Mecamylamine (Active Comparator)
  Interventions: Drug: Mecamylamine
- Control, Varenicline (Active Comparator)
  Interventions: Drug: Varenicline
- Control, placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mecamylamine — A single dose of 10 mg of mecamylamine (via two 5 mg capsules) is given at the start of the mecamylamine arm of the study. This is the only administration of mecamylamine given during the course of the study. Participants' blood pressure and vitals are checked regularly for five hours after drug administration for monitoring and safety assurance.
  Other Names: Inversine
  Arms: Control, Mecamylamine; Schizophrenia, Mecamylamine
Drug: Varenicline — A single dose of 1 mg of varenicline (via two 0.5 mg capsules) is given at the start of the varenicline arm of the study. This is the only administration of varenicline given during the course of the study. Participants' blood pressure and vitals are checked regularly for five hours after drug administration for monitoring and safety assurance.
  Other Names: Chantix
  Arms: Control, Varenicline; Schizophrenia, Varenicline
Drug: Placebo — The placebo contains no active medication. The placebo dose is given via two capsules at the start of the placebo arm of the study. Participants' blood pressure and vitals are checked regularly for five hours after drug administration for monitoring and safety assurance. The placebo has no effects that last for any duration of time.
  Arms: Control, placebo; Schizophrenia, Placebo

SUMMARY:
We are conducting this study to find out if blocking or partially stimulating the effects of nicotine in the brain can affect memory and concentration. Nicotine is the addictive drug found in tobacco products. Our subjects will be people with and without mental illness (schizophrenia), smokers and non-smokers.

We will use a medication called mecamylamine (Inversine) to block the effects of nicotine on the brains of our subjects. We will also use a medication called varenicline (Chantix) to partially increase the effects of nicotine on the brains of our subjects. This study also uses a placebo, a pill that does not have any active ingredients but looks exactly like the mecamylamine and varenicline pills. We will compare the effects of giving mecamylamine or placebo to people who have schizophrenia and people who do not have schizophrenia.

We know that people with schizophrenia smoke heavily and find it harder to stop smoking than most other people do. Studies have shown that people with schizophrenia may smoke more because nicotine helps their concentration and memory. We are interested in helping people with schizophrenia smoke less. Mecamylamine blocks the parts of the brain that react to nicotine and varenicline partially stimulates and partially blocks the parts of the brain that react to nicotine. Both medications may decrease the effects that smoking has on the body.

DETAILED DESCRIPTION:
Taking part in this study will involve one Screening Visit and four Study Visits, all of which will take part over a period of about 3-5 weeks.

SCREENING VISIT We will ask you to come to the Freedom Trail Clinic of Massachusetts General Hospital for a Screening Visit. If you agree to take part in the study, a member of the study staff will explain the study to you and ask you to sign a consent form. You will then have an interview with a study staff member.

We will ask you questions about your current and past mental health and any symptoms you have experienced, such as hearing voices. We will ask you about previous smoking and your current medications. We will review your medical record for psychiatric diagnosis and treatment. Although we hope you will answer all the questions we ask, you may skip over any you choose not to answer. Your answers will be kept confidential.

We will also give you a physical examination. A doctor will fully examine you, including listening to your heart and lungs and feeling your abdomen (belly area). We will also weigh you and take your blood pressure and pulse.

We will need to take a sample of your breath to check for recent smoking. We take this sample by asking you to breathe into a small, hand-held machine. This machine measures a gas in your breath (carbon monoxide) and tells us how much you smoke.

We will ask you for a saliva sample, to check for the use of nicotine and commonly used street drugs, such as marijuana, cocaine, PCP, opiates or amphetamines. We do this by asking you to put a small sponge in your mouth. The sponge soaks up a small sample of saliva. If you test positive for any of these street drugs, you will not be able to take part in the study. The results of the saliva test will not become part of your medical record, but will be recorded in the study records.

If you qualify for the study, we will arrange a date and time for you to return for the first of four study visits. The four visits will be separated by approximately one week. You will continue to take all your regular medications during this study, unless instructed otherwise by a study physician.

FIRST STUDY VISIT The first visit will last about 2½ hours in total. At this visit, you will practice the computer tasks included in the study until you are comfortable with them. These tasks measure your concentration and memory. You do not need to know how to use a computer to do these tasks. They will take about 1½ hours in total to finish.

In one task, we will ask you to watch the screen very closely and press a button every time you see a certain combination of numbers. In another task, we will ask you to remember a letter or word and press the button when you see it again. In another task, you will need to remember the location of a cross and indicate to the location after a period of time. In another task, we will ask you to read words or colors off of a card.

We will also ask you to fill out some questionnaires about your mood and other psychiatric symptoms. These questionnaires take about 20-30 minutes to complete. Although we hope you will answer all the questions, you may skip over any questions that you don't choose to answer. Your answers will be kept confidential. These questionnaires are labeled with a number, and your name does not appear on them. The code that links numbers to names is kept in a locked cabinet in a different location. Your initials will appear on questionnaires.

During the computer tasks, you will be allowed to take smoking breaks or rest breaks if you need to.

TAKING THE STUDY DRUG OR PLACEBO You will receive mecamylamine one time, varenicline one time, and placebo one time during the course of this study, but on different study days. At the second, third, and fourth visits, you will take one of the study drugs or the placebo, but not both. The order in which you take the medication or placebo will be assigned by chance, like the flip of a coin. Neither study staff nor you will know if you have received medication or placebo, although we can find this out in an emergency.

SECOND, THIRD AND FOURTH STUDY VISITS At these next three study visits, we will ask you to take a pill that either contains mecamylamine (10 mg), varenicline (1 mg), or placebo (no active medications). Prior to giving you the pill, we will again ask for a saliva sample to test for nicotine and commonly used street drugs. You will then relax and watch a movie for three hours. We will provide a selection of DVDs for you to choose from and ask that you choose from among this selection. We will provide food, drinks, and snacks, and you will have a comfortable room to sit in. If you prefer to bring your own food, you may do that as well. During this time we will take your blood pressure and pulse every 30 minutes and ask you to fill out a standard questionnaire that asks about side effects that will take 1-2 minutes.

After 3 hours, we will ask you to provide 3 tablespoons of your blood so that we can measure the amount of study medication in your blood. We will destroy your blood sample at the end of the study. You may choose not to have your blood drawn, and you may still participate in the study.

We will then ask you to complete the same tests and questionnaires that you did during the first study visit, and one additional task in which you will be able to earn extra money during each visit. This additional test is a game on the computer called the "face game."

These computer tasks and questionnaires will take about 2 to 2 ½ hours in total to complete. During this time, you will be able to take breaks to relax or smoke between tasks if needed.

ADDITIONAL TASK AT THE END OF THE SECOND STUDY VISIT ONLY During the second visit after the completion of the normal study tasks, we will ask you to do one additional task, which gives you the opportunity to win money. In this task we will ask you to sort cards into three different piles. You will be given the money you have won as you leave the research center that day.

ELIGIBILITY:
Inclusion Criteria for Patients with Schizophrenia:

* Males or females ages 18-68
* Axis I diagnosis of schizophrenia or schizoaffective disorder
* Smoking or Non-smoking
* Negative salivary screen for drugs of abuse
* Stable psychiatric treatment for 4 weeks

Exclusion Criteria for Patients with Schizophrenia

* Current (within the last 6 months) DSM-IV diagnosis of bipolar disorder, PTSD, organic mental disorder, or anorexia nervosa
* Substance use disorder other than nicotine or caffeine in the past 6 months
* Orthostatic blood pressure changes at 3 minutes of > 20 mm Hg systolic or 10 mm Hg diastolic
* Blood Pressure: Women under 50 years of age: Supine baseline systolic blood pressure < 90 mm Hg; Men under 50 years of age: Supine baseline systolic blood pressure < 100 mm Hg; Women and men over 50 years of age: Supine baseline systolic blood pressure < 110 mm Hg
* History of angina, MI within the past 2 years, CHF with LVEF < 40%
* History of syncope or neurocardiogenic syncope
* History of stroke or TIA's
* Glaucoma
* Pyloric Stenosis
* Current pregnancy or lactation
* Renal Insufficiency/Uremia
* Known allergy to mecamylamine
* Inability to give informed consent
* Cognitive impairment secondary to head injury, dementia, general medical condition, or mental retardation
* Current use of antibiotics or sulfa drugs, vasodilators such as alpha blocking agents and nitrates
* Use of investigational medication or device within one month of randomization
* Chronic use of antihypertensive drugs, including diuretics, will be considered on an individual basis

Inclusion Criteria for Healthy Controls:

* Males or females ages 18-68
* Smoking or Non-smoking
* Negative salivary screen for drugs of abuse

Exclusion Criteria for Healthy Controls:

* Current or lifetime Axis I DSM-IV diagnosis or family history of schizophrenia, schizoaffective disorder, or bipolar disorder
* Current (within past 6 months) Axis I DSM-IV diagnosis of major depressive disorder, eating disorder, generalized anxiety disorder or PTSD
* Substance use disorder other than nicotine or caffeine in the past 6 months
* Orthostatic blood pressure changes at 3 minutes of > 20 mm Hg systolic or 10 mm Hg diastolic
* Blood Pressure: Women under 50 years of age: Supine baseline systolic blood pressure < 90 mm Hg; Men under 50 years of age: Supine baseline systolic blood pressure < 100 mm Hg; Women and men over the age of 50: Supine baseline systolic blood pressure < 110 mm Hg
* History of angina, MI within the past 2 years, CHF with LVEF < 40%
* History of syncope or neurocardiogenic syncope
* History of stroke or TIA's
* Glaucoma
* Pyloric Stenosis
* Current pregnancy or lactation
* Renal Insufficiency/Uremia
* Known allergy to mecamylamine
* Inability to give informed consent
* Cognitive impairment secondary to head injury, dementia, general medical condition, or mental retardation
* Current use of antibiotics or sulfa drugs, vasodilators such as alpha blocking agents and nitrates
* Use of investigational medication or device within one month of randomization
* Chronic use of antihypertensive drugs, including diuretics, will be considered on an individual basis

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital; Catherine Fullerton, M.D., M.P.H., Study Director — Massachusetts General Hospital
Locations (1):
- Freedom Trail Clinic, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Roh S, Hoeppner SS, Schoenfeld D, Fullerton CA, Stoeckel LE, Evins AE. Acute effects of mecamylamine and varenicline on cognitive performance in non-smokers with and without schizophrenia. Psychopharmacology (Berl). 2014 Feb;231(4):765-75. doi: 10.1007/s00213-013-3286-3. Epub 2013 Oct 11. PMID 24114425

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were stable, outpatient, non-smokers with schizophrenia on a stable dose of antipsychotic medication for at least 4 wks, from an urban community mental health clinic in Boston. Controls were recruited through media advertisements in the greater Boston area and had no lifetime history of Axis I disorders by SCID
Pre-assignment Details: 89 participants were enrolled, 71 participants (30 patients, 41 controls) completed at least one medication visit and were included in the analyses. 4 participants (3 with schizophrenia, 1 control) missed one and 5 participants (3 with schizophrenia, 2 controls) missed 2 of the 3 medication visits.
Groups:
- Schizoph: Mecamylamine (Wk1),Varenicline (Wk2), Placebo (Wk3); Control: Mecamylamine (Wk1),Varenicline (Wk2), Placebo (Wk3): Mecamylamine: A single dose of 10 mg of mecamylamine (via two 5 mg capsules) is given at the start of the mecamylamine arm of the study. This is the only administration of mecamylamine given during the course of the study. Participants' blood pressure and vitals are checked regularly for five hours after drug administration for monitoring and safety assurance.
- Schizoph: Placebo (Wk1), Mecamylamine (Wk2), Varenicline (Wk3); Control: Placebo (Wk1), Mecamylamine (Wk2), Varenicline (Wk3): Varenicline: A single dose of 1 mg of varenicline (via two 0.5 mg capsules) is given at the start of the varenicline arm of the study. This is the only administration of varenicline given during the course of the study. Participants' blood pressure and vitals are checked regularly for five hours after drug administration for monitoring and safety assurance.
- Schizoph: Varenicline (Wk1), Placebo (Wk2), Mecamylamine (Wk3); Control: Varenicline (Wk1), Placebo (Wk2), Mecamylamine (Wk3): Placebo: The placebo contains no active medication. The placebo dose is given via two capsules at the start of the placebo arm of the study. Participants' blood pressure and vitals are checked regularly for five hours after drug administration for monitoring and safety assurance. The placebo has no effects that last for any duration of time.
Period: Week 1
Arm/Group | Schizoph: Mecamylamine (Wk1),Varenicline (Wk2), Placebo (Wk3) | Schizoph: Placebo (Wk1), Mecamylamine (Wk2), Varenicline (Wk3) | Schizoph: Varenicline (Wk1), Placebo (Wk2), Mecamylamine (Wk3) | Control: Mecamylamine (Wk1),Varenicline (Wk2), Placebo (Wk3) | Control: Placebo (Wk1), Mecamylamine (Wk2), Varenicline (Wk3) | Control: Varenicline (Wk1), Placebo (Wk2), Mecamylamine (Wk3)
Started | 10 | 10 | 10 | 14 | 14 | 13
Completed | 10 | 10 | 10 | 14 | 14 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 2
Arm/Group | Schizoph: Mecamylamine (Wk1),Varenicline (Wk2), Placebo (Wk3) | Schizoph: Placebo (Wk1), Mecamylamine (Wk2), Varenicline (Wk3) | Schizoph: Varenicline (Wk1), Placebo (Wk2), Mecamylamine (Wk3) | Control: Mecamylamine (Wk1),Varenicline (Wk2), Placebo (Wk3) | Control: Placebo (Wk1), Mecamylamine (Wk2), Varenicline (Wk3) | Control: Varenicline (Wk1), Placebo (Wk2), Mecamylamine (Wk3)
Started | 10 | 10 | 10 | 14 | 14 | 13
Completed | 10 | 10 | 10 | 14 | 14 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 3
Arm/Group | Schizoph: Mecamylamine (Wk1),Varenicline (Wk2), Placebo (Wk3) | Schizoph: Placebo (Wk1), Mecamylamine (Wk2), Varenicline (Wk3) | Schizoph: Varenicline (Wk1), Placebo (Wk2), Mecamylamine (Wk3) | Control: Mecamylamine (Wk1),Varenicline (Wk2), Placebo (Wk3) | Control: Placebo (Wk1), Mecamylamine (Wk2), Varenicline (Wk3) | Control: Varenicline (Wk1), Placebo (Wk2), Mecamylamine (Wk3)
Started | 10 | 10 | 10 | 14 | 14 | 13
Completed | 10 | 10 | 10 | 14 | 14 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eighty-nine participants were enrolled, and 71 participants (30 patients, 41 controls) completed at least one medication visit and were included in the analyses. Four participants (3 with schizophrenia, 1 control) missed one and 5 participants (3 with schizophrenia, 2 controls) missed two of the three medication visits.
Groups:
- Schizophrenia: Study participants in the schizophrenia group were clinically stable, outpatient, non-smokers with schizophrenia on a stable, clinically determined dose of antipsychotic medication for at least 4 weeks, which were recruited from an urban community mental health clinic in Boston. Diagnoses were confirmed by clinical interview and medical record review
- Control: Healthy volunteers were recruited through media advertisements in the greater Boston area and had no lifetime history of Axis I disorders by SCID interview and no firstdegree relatives with Axis I disorders by history
- Total: Total of all reporting groups
Arm/Group | Schizophrenia | Control | Total
Number analyzed (Participants) | 30 | 41 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10) | 37 (16) | 42 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 23 | 33
  Male | 20 | 18 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 24 | 22 | 46
  African American | 5 | 12 | 17
  Asian or Pacific Islander | 0 | 4 | 4
  Unknown | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 30 | 41 | 71

OUTCOME MEASURES:

1. Primary Outcome: Effects of Mecamylamine and Varenicline Compared With Placebo in Schizophrenia and Control Groups on Prolonged Attention as Assessed With the CPT-IP Hit Reaction Time Variability
Description: The Continuous Performance Test-Identical Pairs, CPT-IP, Version 4.0 was developed and normed for use in people with schizophrenia and normal controls. This task estimates attention by requiring an individual to push a response key when two identical pairs of shapes or numbers are presented in sequence. Stimuli were presented with increasing cognitive load: 2-, 3-, and 4-digit targets. Outcome variables measured included correct hits, hit reaction time (HRT), errors of commission: false alarms and random errors, and the primary outcome, variability, or standard deviation, of hit reaction time, HRT-SD. There is only one outcome measure time point because cognitive outcomes were analyzed using crossover analyses of covariance (ANCOVA) with drug (mecamylamine vs. varenicline vs. placebo) as a within subject factor, diagnosis (schizophrenia vs. control) as a between subject factor, as well as study period and drug administration sequence as between subject crossover design factors.
Time Frame: Baseline (week 0), week 1, week 2 and week 3 as one time point (see outcome measure description)
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Schizophrenia: Mecamylamine; Control: Mecamylamine: Mecamylamine: A single dose of 10 mg of mecamylamine (via two 5 mg capsules) is given at the start of the mecamylamine arm of the study. This is the only administration of mecamylamine given during the course of the study. Participants' blood pressure and vitals are checked regularly for five hours after drug administration for monitoring and safety assurance.
- Schizophrenia: Varenicline; Control: Varenicline: Varenicline: A single dose of 1 mg of varenicline (via two 0.5 mg capsules) is given at the start of the varenicline arm of the study. This is the only administration of varenicline given during the course of the study. Participants' blood pressure and vitals are checked regularly for five hours after drug administration for monitoring and safety assurance.
- Schizophrenia: Placebo; Control: Placebo: Placebo: The placebo contains no active medication. The placebo dose is given via two capsules at the start of the placebo arm of the study. Participants' blood pressure and vitals are checked regularly for five hours after drug administration for monitoring and safety assurance. The placebo has no effects that last for any duration of time.
Arm/Group | Schizophrenia: Mecamylamine | Schizophrenia: Varenicline | Schizophrenia: Placebo | Control: Mecamylamine | Control: Varenicline | Control: Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 41 | 41 | 41
ms | 141.6 (57.5) | 120.5 (58.5) | 123.1 (44.9) | 91.2 (31.1) | 83.2 (30.2) | 87.8 (21.7)

2. Secondary Outcome: Effects of Mecamylamine and Varenicline Compared With Placebo in Schizophrenia and Control Groups on Cognitive Interference as Assessed by The Three-card Stroop Task
Description: In the 3-card Stroop Task, 3 cards were presented; the 1st contained color names printed in black ink, the 2nd contained colored patches of ink, the 3rd contained color names printed in incongruously colored ink. Participants were asked to read or name as many items as possible in 45 seconds for each condition. Individuals are asked to identify the color of the ink of a word. They may be distracted by the presence of a word that states another color (i.e. the word "blue" written in green ink would require the answer green).The interference score was calculated by dividing the color-word score by the color score. There is only one outcome measure time point because cognitive outcomes were analyzed using crossover analyses of covariance (ANCOVA) with drug (mecamylamine vs varenicline vs pbo) as a within subject factor, diagnosis (schizophrenia vs. control) as a between subject factor as well as study period and drug administration sequence as between subject crossover design factors
Time Frame: Baseline (week 1), week 2, week 3, week 4 analyzed as a single time point
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Schizophrenia: Mecamylamine | Schizophrenia: Varenicline | Schizophrenia: Placebo | Control: Mecamylamine | Control: Varenicline | Control: Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 41 | 41 | 41
score | 50.2 (6.8) | 52.8 (8.0) | 50.3 (8.3) | 54.4 (10.5) | 53.3 (9.2) | 53.5 (8.6)

3. Secondary Outcome: Effects of Mecamylamine and Varenicline Compared With Placebo in Schizophrenia and Control Groups on Sustained Attention as Assessed by The N-back Task
Description: The N-back task with 1- and 2-back parametric conditions was used. During the task, a letter was displayed for 1,500 ms every 2 s with a 500 ms isi. Participants were asked to press the "1" key for letters that corresponded to the letter 1 back for the 1-back condition, the "2" key for the 2-back condition, and the "3" key for nontarget letters. Outcome variable presented is hit reaction time There is only one outcome measure time point because this outcome was analyzed using crossover analyses of covariance (ANCOVA) with drug (mecamylamine vs. varenicline vs. placebo) as a within subject factor, diagnosis (schizophrenia vs. control) as a between subject factor, as well as study period and drug administration sequence as between subject crossover design factors.
Time Frame: Baseline (week 1), week 2, week 3, week 4 analyzed as a single time point
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Schizophrenia: Mecamylamine | Schizophrenia: Varenicline | Schizophrenia: Placebo | Control: Mecamylamine | Control: Varenicline | Control: Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 41 | 41 | 41
ms | 909.2 (250.9) | 931.2 (297.9) | 894.4 (282.1) | 864.6 (253.9) | 795.8 (241.7) | 827.5 (229.3)

4. Secondary Outcome: Effects of Mecamylamine and Varenicline Compared With Placebo in Schizophrenia and Control Groups on Working Memory as Assessed by The Visual Spatial Working Memory (VSWM) Task
Description: In the Visual spatial working memory (VSWM), participants were asked to place the cursor where the symbol appeared immediately after its display. For 16 additional trials, participants were asked to identify the symbol location after a 30-second delay. During the delay, participants were distracted by being asked to read aloud words appearing on the screen at 2-second intervals. The outcome of interest in this task were the average distance from the target for immediate and delayed recall There is only one outcome measure time frame because this outcome was analyzed using crossover analyses of covariance (ANCOVA) with drug (mecamylamine vs. varenicline vs. placebo) as a within subject factor, diagnosis (schizophrenia vs. control) as a between subject factor, as well as study period and drug administration sequence as between subject crossover design factors.
Time Frame: Baseline (week 1), week 2, week 3, week 4 analyzed as a single time point
Measure: Mean (Standard Deviation); unit: Distance (in)
Arm/Group | Schizophrenia: Mecamylamine | Schizophrenia: Varenicline | Schizophrenia: Placebo | Control: Mecamylamine | Control: Varenicline | Control: Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 41 | 41 | 41
Distance (in) | 2.83 (0.71) | 2.72 (0.66) | 2.87 (0.76) | 2.29 (0.54) | 2.28 (0.54) | 2.25 (0.53)

ADVERSE EVENTS:
Arm/Group | Schizophrenia | Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/41
Other Adverse Events (participants affected / at risk) | 0/30 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No